CLINICAL TRIAL: NCT05213819
Title: Additional Contribution of Phonophoresis and Low-Level Laser Therapy to Exercise in the Treatment of Carpal Tunnel Syndrome by Clinical, Electrophysiological and Ultrasonographical Evaluation
Brief Title: Phonophoresis, Low-Level Laser Therapy and Exercise in the Treatment of Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Nazlı Karaman, MD, Principal Investigator, Kutahya Health Sciences University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCakil1
Record Dates: First submitted 2021-12-28; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal tunnel syndrome; Phonophoresis; Low-Level Laser Therapy; Exercise; Electrophysiological; Ultrasonographical
MeSH Terms: conditions — Carpal Tunnel Syndrome; Motor Activity

ARMS (1):
- Carpal tunnel syndrome (Other): Patients with carpal tunnel syndrome were treated with phonophoresis, low level laser therapy and exercise.
  Interventions: Other: Carpal Tunnel Syndrome

INTERVENTIONS:
Other: Carpal Tunnel Syndrome

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common peripheral nerve compression syndrome. There is insufficient evidence about the efficacy and superiority of conservative treatment methods. The purpose of this study was to evaluate the additional contribution of phonophoresis and Low-Level Laser Therapy (LLLT) to exercise in patients with the CTS.

Study design: A single-blind randomized controlled study. Methods: Forty-five patients with clinical and electrophysiologic evidence of moderate CTS were included in the study. The patients were randomized into three groups. Group 1 received phonophoresis and exercise, group 2 received LLLT and exercise and group 3 received exercise alone. All patients were evaluated electrophysiologically, clinically and ultrasonographically before treatment and 6th and 12th week after the treatment.

DETAILED DESCRIPTION:
45 patients in total (5 males, 40 females; mean age 50.2±10.0 years; ranged 26 to 69 years) having clinical and electrophysiologic findings of moderate CTS were examined. Inclusion criteria were as follows: age older than 18 years, positive Tinel's sign or positive Phalen's sign, pain or paresthesia in the median nerve course, pain or paresthesia aggravated at night and moderate CTS according to the American Association of Electrodiagnostic Medicine (AAEM) guidelines (10,11). Exclusion criteria were as follows: metabolic diseases (including diabetes mellitus, thyroid and chronic kidney diseases), rheumatoid arthritis, wrist trauma, pregnancy, corticosteroid treatment in the last 3 months, physical or medical treatment in the last month. The participants were randomly categorized into three groups with an indiscriminate number table as Group 1 (phonophoresis combined with exercise, n:15), Group 2 (LLLT combined with exercise, n:15) and Group 3 (exercise only, n:15).

Phonophoresis was administered to the course of carpal tunnel for 8 minutesfor every session at 3 MHz frequency and 1.0 W/cm2 intensity, pulsed mode (1:4) ultrasound having a transducer having a surface area of 1.4 cm2 (Sonicator 730, Metler Electronics, USA). Ketoprophen %2.5 gel was used. Patients underwent this therapy 5 days a week, for 3 weeks.

A Gal-Al-As diode laser device (Endolaser 476, Enraf Nonius, Hollanda) was the LLLT source having 30 mW power output and 830 nm wavelength. The probe irradiated 3 points in total on the volar side at the wrist. A one minute irradiation per point (3 minutes in total) was determined as the single dose of irradiation. The dose for every tender joint was 1.8 joule. The total and acculumated doses after 15 treatments were 5.4 and 81 joules, respectively. This therapy was applied 5 days a week, for 3 weeks.

All the individuals were asked to complete nerve and tendon gliding activities of Totten and Hunter (12). In addition, a book letex plaining the activities was provided to all individuals. Patients were called by phone weekly and they were checked and reminded about their exercises. For tendon gliding exercises, the fingers were formed into five seperate positions, as straight, hook, fist, table top, and straight fist. For the median nerve-gliding exercising, putting the hand and wrist in six seperate positions caused the mobilization of the median nerve. The neck and the shoulder were in a neutral position, and the elbow in supination and 90 degrees flexion over all these exercises. Each seperate position was uphold for 5 seconds. The exercising wasrepeated as five sessions every day. 10 repetitions of each exercising was made for every session, and exercise therapy lasted for 3 weeks.

Data including age, gender, body mass index (BMI) and disease duration (months) were recorded for all patients on admission.The most symptomatic hand was included in patients with bilateral CTS. Pain intensity in the rest and activity wasassessed by the visual analog scale (VAS), which the individuals could specify the pain evaulationon a 10 cm distance, between 0 (no pain) and 10 (the most intense pain).

The Boston Carpal Tunnel Questionnaire (BCTQ) is self-applied and assesses the symptom severity and functional status in CTS patients (13). BCTQ is including two subscales. The Boston Symptom Severity Scale (BSSS) consists of 11 questions and the Boston Functional Status Scale (BFSS) 8 questions. Each question is assessed on a 1-point (mildest pain) to 5-point (most intense pain) scoring system. The each scale's scoring was determined as the average of all items. Sezgin et al (14) has been validated the Turkish version of BCTQ.

Electrophysiologic examinations of all patients were performed at 22-24 °C room temperature using a 2-channel Dantec Keypoint Portable model electromyography (EMG) device of Alpine Biomed Company (Natus Medical Incorporated Corporate Headquarters 1501 Industrial Road San Carlos, CA 94070 USA). The band-pass filter was 20 Hz to 3 kHz, sweep speed velocity 2 ms/division, and gain 10 lV/division. Electrophysiological studies were performed according to the AAEM guidelines (10,11). The studies included an electromyographic investigation of the muscles of abductor pollicis brevis, adductor digiti minimi and ﬂexor carpi radialis, and the median and ulnar nerves'motor and antidromic sensorial conduction velocities. In order to diagnose CTS, the electrophysiological criteria was determined as median nerve's distal motor latency of >4.2 ms from the wrist to abductor pollicis brevis, and the seperation between the median and ulnar sensorial distal latencies surpassing 0.5 ms.

CTS was categorized electrodiagnostically per the following criteria (15). 1- Mild CTS: Elongation (absolute or relative) and/or decrease in sensory action potential (SNAP) amplitude in sensory or mixed distal latency (DL) (orthodromic, antidromic, or palmar). 2- Moderate CTS: In addition to the above, elongation in the median motor DL. 3- Severe CTS: Together with the prolongation of median motor and sensory latencies, failure to obtain sensory or mixed action potentials or low amplitude compound muscle action potential (CMAP) or failure to obtain it, fibrillations, attenuation in full twitching in needle EMG, observing changes in motor unit potentials. Moderate CTS patients diagnosed by electrophysiological findings were included in the research.

Ultrasonographic studies were implemented using high-resolution US having a 12-3 MHz linear array transducer (Philips HDI Envisor; Philips Medical Systems, Bothell, WA, USA). The evaluations were made as all wrists in the neutral position as the palm being up and the ﬁngers semi-extended. The median nerve'sfull course was determined within the carpal tunnel in the transverse and sagittal planes. The median nerve'scross-sectional area (CSA), transverse and anteroposterior diameters were evaluated at the pisiform bone level of proximal carpal tunnel, and its CSA was determined by a tracking approach in which the median nerve'smargin was quantified using electronic caliper. Distal carpal tunnel was not used for any measurements (16). Three measurement repetitions were made and the average of these values was determined for every wrist. The transverse diameter was divided by anterio-posterior diameter and the flattening ratio (FR) was calculated.

The researchers assessed ultrasonographic, electrodiagnostic and clinical examinations were blinded to assigned therapies and to each other. The same researchers determined all these parameters once again at the 6th and 12th weeks after the initiation.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years
* positive Tinel's sign or positive Phalen's sign
* pain or paresthesia in the median nerve course
* pain or paresthesia aggravated at night
* moderate CTS according to the American Association of Electrodiagnostic Medicine (AAEM) guidelines

Exclusion Criteria:

* metabolic diseases (including diabetes mellitus, thyroid and chronic kidney diseases)
* rheumatoid arthritis
* wrist trauma
* pregnancy
* corticosteroid treatment in the last 3 months
* physical or medical treatment in the last month

Ages: 26 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-02-20 (Actual); Primary Completion 2015-02-20 (Actual); Study Completion 2015-02-20 (Actual)

PRIMARY OUTCOMES:
Body mass index | 12 weeks
  kg/m2

SECONDARY OUTCOMES:
Duration of disease | 12 weeks
  months
Sex | 12 weeks
  female, male
The Boston Carpal Tunnel Questionnaire | 12 weeks
  Boston symptom severity scale and Boston functional status scale
visual analog scale (VAS) | 12 weeks
  visual analog scale at rest and visual analog scale on activity
Ultrasonographic parameters | 12 weeks
  cross-sectional area, flattening ratio
Electrophysiologic parameters | 12 weeks
  motor distal latancy, motor amplitude,sensory nerve velocity, sensory distal latancy,sensory amplitude

CONTACTS AND LOCATIONS:
Overall Officials: Nazlı Karaman, Principal Investigator — Kütahya Health Sciences University
Locations (1):
- Health Sciences University, Evliya Çelebi Training and Research Hospital, Kütahya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes